CLINICAL TRIAL: NCT04453098
Title: Results at 10 Years of the RESOLVE Study (REverse Metabolic SyndrOme by Lifestyle and Various Exercise)
Brief Title: Results at 10 Years of the RESOLVE Study (RESOLVE+10)
Acronym: RESOLVE+10
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital CHU Clermont-Ferrand, 58 rue Montalembert 63003 Clermont-Ferrand, France (Unknown); Université d'Auvergne (Other); LaPSCo laboratory, Physiological and Psychosocial Stress" team, UMR CNRS 6024, Clermont-Ferrand, France (Unknown); LaPEC laboratory (EA 4278), University of Avignon, Avignon, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AOI 2018 DUTHEIL; 2019-A01016-51 (Other: ANSM)
Record Dates: First submitted 2020-06-22; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Metabolic Syndrome
Keywords: physical activity; spa residential lifestyle program; prevention
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity | interventions — Diet

STUDY DESIGN:
Intervention Model Description: participants receive an intervention throughout the protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Re group (Experimental): high-Resistance-moderate-endurance, participants performed 10 repetitions at 70% of one maximal repetition in resistance and 30% of VO2-peak for endurance training
  Interventions: Behavioral: 3-week residential program based on a tryptic (diet,
- rE group (Experimental): moderate-resistance (30%) - high-Endurance (70%)
  Interventions: Behavioral: 3-week residential program based on a tryptic (diet,
- re group (Experimental): moderate-resistance (30%) - moderate-endurance (30%).
  Interventions: Behavioral: 3-week residential program based on a tryptic (diet,
- control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: 3-week residential program based on a tryptic (diet, — 3-week residential program based on a tryptic (diet, exercise, education). The three weeks intervention was followed by a 1-year at-home follow-up.
  In the original protocol, participants were involved in a 3-week residential program based on a tryptic (diet, exercise, education).
  Arms: Re group; rE group; re group

SUMMARY:
10-year effect of a lifestyle intervention program (exercise, sedentary lifestyle and dietary diet) on abdominal visceral adipose tissue (primary endpoint of the RESOLVE study 10 years ago): influence of kinetics abdominal visceral adipose tissue loss in the first year of follow-up on abdominal visceral adipose tissue at 10 years

DETAILED DESCRIPTION:
The RESOLVE + 10 protocol was design to provide a 10-year effect of a lifestyle intervention program (exercise, sedentary lifestyle and dietary diet) on abdominal visceral adipose tissue.

In the present protocol, parameters are measured just once, during 3 hours, to compared the results with those of the protocol RESOLVE (5 measurement times over a year 10 years ago: before the thermal modification program of the lifestyle ( exercise, sedentary lifestyle and diet) of 3 weeks (D0), after the thermal program (D21), at the 3rd month (M3), 6th month (M6) and 12th month of follow-up (M12), to which was matched a healthy control group).

Statistical analysis will be performed using Stata software (version 13; Stata-Corp, College Station, Tex., USA). All statistical tests will be two-sided and p inferior to 0.05 will be considered significant. Qualitative variables will be described in terms of numbers and proportions. Quantitative variables will be described in terms of numbers, mean standard deviation or median according to statistical distribution (normality studied using Shapiro-Wilk test). Graphic representations will be complete presentations of results. Comparisons between patients and controls, concerning loss of abdominal visceral adipose tissue at 10 years, will be performed using Student t-test or Mann-Whitney test if the assumptions of anova are not met (normality and homoscedasticity analyzed using Fisher-Snedecor test). The results will be expressed as effect-size and 95 percent confidence intervals. The primary analysis should be completed by multivariable analysis (linear regression with logarithmic transformation of dependent outcome if necessary) considering an adjustment on covariates fixed according to univariate results and clinical relevance. The results will be expressed as regression coefficients and 95percent confidence intervals. Furthermore, the abdominal visceral adipose tissue loss kinetics in the first year of follow-up will be considered an independent variable and treated as a functional variable. The intra-group comparisons (for patients and for controls) will be performed using paired statistical tests: paired t-test or Wilcoxon test. The results will be expressed as effect-size and 95 percent confidence intervals. Comparisons between independent groups will be done similarly as presented previously for other quantitative outcomes (body composition, quality of life, skin conductance, etc.). Multivariable analyses will be applied similarly as described previously. The comparisons concerning categorical variables will be realized using Chi-squared or when appropriate Fischer-exact test. The relations between quantitative outcomes will be analyzed using correlation coefficients (Pearson or Spearman according to statistical distribution). Considering the several multiple comparisons, a correction of the type I error will be applied (Sidak's correction).

ELIGIBILITY:
Inclusion Criteria:

* patients and healthy controls included in the RESOLVE study

Exclusion Criteria:

* refusal of participation

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Abdominal visceral adipose tissue loss, a primary cardiovascular risk (CVR) factor, highly related to morbidity and mortality | Year 10
  to assess the ability of a lifestyle program in decreasing abdominal visceral fat, one of the major health-related factor It will be assessed from dual-energy X-ray absorptiometry

SECONDARY OUTCOMES:
weight | Year 10
  measured in kilogramms
systolic blood pressure | Year 10
  measured in millimeter of mercure
diastolic blood pressure | Year 10
  measured in millimeter of mercure
Waist circumference | Year 10
  measured in centimeter
heart rate | Year 10
  measured in battment per minutes
Muscle mass | Year 10
  measured using Impedancemeter, Densitometry x-ray absorption, Peripheral quantitative computed tomography (pQCT) and Quantitative ultrasounds (QUS)
fat mass | Year 10
  measured using Impedancemeter, Densitometry x-ray absorption, Peripheral quantitative computed tomography (pQCT) and Quantitative ultrasounds (QUS)
bone structure | Year 10
  measured using Impedancemeter, Densitometry x-ray absorption, Peripheral quantitative computed tomography (pQCT) and Quantitative ultrasounds (QUS)
Epicardial adipose tissue | Year 10
  measures of epicardial adipose tissue using Magnetic resonance imaging (MRI) and echocardiography
myocardial triglycerides | Year 10
  measures of myocardial triglycerides using MRI
cardiac remodeling and function | Year 10
  measures cardiac remodeling and function using MRI and echocardiography)
Depression | Year 10
  Assessing depression using Hospital anxiety and depression scale- HAD. It's a 14-item questionnaire about frequency of perception about anxious (HAD-A: 7 items) and depressive (HAD-D: 7 items) symptoms. Items are made of a 4-point scale frequency of symptoms, varying from "never" to "always". Scores higher than 8 for HAD-A or HAD-D mean a possible symptomatology, and scores higher than 11 mean a clear and proper diagnostic of depressive or anxious disorder.
anxiety | Year 10
  Assessing anxiety using State and trait anxiety inventory which consists of separate self-report scales measuring to distinct anxiety concepts: state anxiety and trait anxiety. Both state and trait anxiety are explored by a 20-item questionnaire made of a 4-point scale from "never" to "always".
General health | Year 10
  Assessing general health using General Health Questionnaire with 36 items (SF-36)
Stress | Year 10
  Assessing stress using visual analog scale of 100 mm, ranging from very low (0) to very high (100).
Fatigue | Year 10
  Assessing fatigue using visual analog scale of 100 mm, ranging from very low (0) to very high (100).
Sleep | Year 10
  Assessing sleep using visual analog scale of 100 mm, ranging from very low (0) to very high (100).
Burnout | Year 10
  Assessing burnout using Maslach Burnout Inventory, composed of 22 items designed to assess the three components of the burn-out syndrome: emotional exhaustion (9 items), depersonalization (5 items) and reduced personal accomplishment (8 items). Items are made of a 7-point scale frequency of feelings, varying from "never" to "every day". The scores for each component of the burn-out syndrome are considered separately and are not combined into a single total score. If desired for participant feedback, each score can be coded as low, average, or high.
Mindfulness | Year 10
  Assessing mindfulness using Freiburg Mindfulness Inventory a consistent and reliable scale evaluating several important aspects of mindfulness. Mindfulness has been described as a non-elaborative, non-judgmental present-centred awareness in which each thought, feeling or sensation that arises in the attention field is acknowledged and accepted as it is. Mindfulness appears as an attribute of consciousness long believed to promote well-being. Each self-descriptive statement of the FMI is evaluated using a four-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree)
Coping strategy | Year 10
  Assessing coping using Brief COPE Questionnaire made to evaluate self-perceived reaction to a particular situation. The 28 items of the BCQ explore the 14 different theoretically identified coping responses (with two items for each of the measured coping strategies): self-distraction, active coping, denial, substance use, use of emotional support, use of instrumental support, Behavioral disengagement, venting, positive reframing, planning, humor, acceptance, religion, and self-blame. Items of BCQ are scored on a four-point Likert-type scale, ranging from 1 = strongly disagree to 4 = strongly agree.
Emotions | Year 10
  Assessing emotions using Emotion Regulation Questionnaire a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: 1) cognitive reappraisal and 2) expressive suppression. Respondents answer each item on a 7-point
Perception of work | Year 10
  Assessing perception of work using Job Content Questionnaire of Karasek which assessed job demands, job control and social support through 26 items. The questionnaire measures 9 items of job demands, 9 items of job control and 8 items of social support. Items are scored on a four-point Likert-type scale, ranging from 1 = strongly disagree to 4 = strongly agree. Among the 26 items, 5 negative statements require reverse scoring. From French data, the job strain threshold is set for a demands score higher than 20 and a control score lower than 71; the isostrain threshold is determined from a combining score of job strain and social support lower than 24. We would ask the participants to fulfil the questionnaire from memories that they keep of their work.
Self-efficacy | Year 10
  Assessing self-efficacy using Perceived self-efficacy scale created to assess a general sense of perceived self-efficacy with the aim in mind to predict coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events. Responses are made on a 4-point scale for the 10 items (from "false" to "true"). The final composite score (ranged from 10 to 40) is obtained by summing up the responses to all 10 items. An example of item is "I am confident that I could deal efficiently with unexpected events".
Addiction | Year 10
  Assessing addiction to work using Work Addiction Risk test (WART). The WART is a self-administered test with 25 statements for which the answers are scored 1-never true to 4-always true [20,26]. Respondents read the statements and mark their answers to describe their work habits [19,27]. The total score is the sum of the responses to the items-25 to 100-and the higher the score, the more one is considered addicted to work [18,21]. Scores from 25 to 56 were defined as "at low-risk of work addiction"; 57 to 66 as "at medium-risk of work addiction", and from 67 to 100 as "at high-risk of work addiction".
Alexithymia | Year 10
  Assessing alexithymia using Toronto Alexithymia Scale For this scale, a three-factor structure was proposed: difficulty identifying feelings, difficulty describing feelings and externally oriented thinking. Responses are made on a 5-point scale from "strongly agree" to "strongly disagree".
Illness perception | Year 10
  Assessing illness perception using Brief Illness Perception Questionnaire (B-IPQ), adapted for stress at work). It's a self-questionnaire comprising an 11-point scale, including 8 items measuring cognitive and emotional illness perceptions (consequences, timeline, personal control, treatment control, symptoms, coherence, illness concern and negative emotions). The total score is calculated by averaging all items (after reversed some items). A high score meant that diabetes was perceived as a threat.
Metacognition | Year 10
  Assessing metacognition using MetaCognition Questionnaire. It is a 30-item questionnaire made of 5-point scales. The MCQ-30 is structured in five factors: cognitive confidence, positive beliefs about worry, cognitive self-consciousness, negative beliefs about uncontrollability of thoughts and danger, and beliefs about need to control thoughts.
Time perception | Year 10
  Assessing time perception using Zimbardo Time Perspective Inventory, a self-reported questionnaire comprising 56 items. Responses are made on a 5-point scale from "very uncharacteristic" to "very characteristic". It explores 3 temporalities and 5 dimensions.
Life style | Year 10
  Assessing factors regarding lifestyle are related to smoking, alcohol, coffee, food intake (questionnaires), and physical activity (Recent Physical Activity Questionnaire)
Treatment perception | Year 10
  Assessing factors regarding psychology and treatment are related to perception of treatment (Beliefs about Medicines Questionnaire), adherence to treatment (Visual analog scales from never to always), barriers to treatment (QUILAM) and treatment satisfaction (treatment SATisfaction with MEDicines Questionnaire).
questionnaires used 10 years ago | Year 10
  Understanding and knowledge about the metabolic syndrome (4 items), comparative optimism (4 items), motivation to eat healthy (16 items) and motivation to practise physical activity (16 items).
Cholesterol | Year 10
  Blood analyses on HDLc and LDL-cholesterol
HbA1c | Year 10
  Blood analyses on HbA1c
Triglycerides (TG) | Year 10
  Blood analyses on Triglycerides (TG)
Cortisol | Year 10
  Blood analyses on Cortisol
DHEAS | Year 10
  Blood analyses on DHEAS
Leptin | Year 10
  Blood analyses on Leptin
BDnF | Year 10
  Blood analyses on BDnF
Cytokines | Year 10
  Blood analyses on Pro-inflammatory Cytokines: IL-1β, IL-6, IL-1, TNFα, NPY
Telomeres length | Year 10
  Blood analyses on Telomeres length
Genetic polymorphisms related to stress | Year 10
  Polymorphism of the angiotensin converting enzyme and Polymorphism of the serotonin are measured by Blood cells
carotid intima-media thickness | Year 10
  Assessing on carotid intima-media thickness by high-resolution B-mode ultrasound.
blood flow velocity | Year 10
  Assessing on blood flow velocity by laser speckle contrast imaging (LSCI) and microvascular perfusion by laser-doppler flowmetry (LDF), flowmotion and Iontophoresis procedure.
microvascular perfusion | Year 10
  Assessing microvascular perfusion by laser-doppler flowmetry (LDF).
flowmotion | Year 10
  Assessing flowmotion
iontophoresis | Year 10
  Assessing iontophoresis procedure
heart rate variability | Year 10
  Assessing heart rate variability by Holter
skin conductance | Year 10
  Assessing skin conductance by Wristband electrodes - Empatica 4.
Quantification of liver steatosis and fibrosis | Year 10
  Liver steatosis by MRI, fibroscanner (ultrasonic attenuation) and Aixplorer (Lipersonic Imagine®).
Quantification of liver fibrosis | Year 10
  Liver fibrosis by fibroscanner (liver stiffness) and fibrotest
Vo2max | Year 10
  Assessing factors regarding fitness are related to Vo2max (maximal exercise test)
Fitness | Year 10
  Assessing factors regarding fitness are related to 6-minutes walking test.
strength | Year 10
  Assessing factors regarding fitness are related to strength
leptin variation | Year 10
  Blood analyses on leptin
ghrelin variation | Year 10
  Blood analyses on ghrelin
NPY variation | Year 10
  Blood analyses on NPY
adiponectin variation | Year 10
  Blood analyses on adiponectin
Evaluation of CCK level | Year 10
  Blood analyses on CCK
Evaluation of VEGF level | Year 10
  Blood analyses on VEGF
Evaluation of PAI1 level | Year 10
  Blood analyses on PAI1
insulin level | Year 10
  Blood analyses on insulin
HbA1c level | Year 10
  Blood analyses on HbA1c
blood glucose level | Year 10
  Blood analyses on blood glucose
albumin level | Year 10
  Blood analyses on blood albumin
transthyretin level | Year 10
  Blood analyses on transthyretin
Homeostasis | Year 10
  Blood analyses on Homeostasis (Fibroblast growth factor 23)
Osteoresorption | Year 10
  Blood analyses on Osteoresorption (C-terminal Telopeptide of Type I collagen)
Osteoformation | Year 10
  Blood analyses on Osteoformation (decarboxylated osteocalcine and BSAP)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Dutheil, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France